CLINICAL TRIAL: NCT05559619
Title: Effect of Laser Acupuncture on Forearm Bone Mineral Density and Wrist Pain in Osteoporotic Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed M Maged, MD, professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 65
Record Dates: First submitted 2022-09-26; First posted 2022-09-29 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Osteoporosis, Postmenopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Calcium Carbonate; Cholecalciferol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug treatment group (Active Comparator): 34 postmenopausal women who only received oral calcium and vitamin D3 supplement (Calcium D3F® (Arab Company for Pharmaceutical& medicinal plants (MEPACO-MEDIFOOD, EGPYT). Each tablet contains 1000 mg of natural calcium carbonate, 1000 IU vitamin D3 (0.025 mg) and 0.25 mg Sodium Fluoride. They received 1 tablet once daily for 12 weeks
  Interventions: Drug: Calcium carbonate; Drug: Vitamin D3
- Drug treatment + laser acupuncture group (Active Comparator): 34 postmenopausal women who received laser acupuncture therapy in addition to the same calcium and vitamin D3 supplement for 12 weeks.
  Interventions: Drug: Calcium carbonate; Drug: Vitamin D3; Device: laser acupuncture therapy

INTERVENTIONS:
Drug: Calcium carbonate — 1000 mg of natural calcium carbonate once daily for 12 weeks
  Other Names: Calcium D3F
Drug: Vitamin D3 — 1000 IU vitamin D3 once daily for 12 weeks
  Other Names: Calcium D3F
Device: laser acupuncture therapy — The patient was in crock lying for stimulation of acupoints in abdomen and lower limbs then asked to be in side lying for stimulation of acupoints in the back. After disinfection of the skin and careful localization of the acupoints, low level laser therapy (LLLT) (model: Lis 1050, SN: EM 13481014, manufactured by EME srl, Italy) was applied bilaterally on Dazhu (BL 11), Ganshu(BL 18), Pishu (BL20), Shenshu (BL23), Zusanli (ST 36), Sanyinjiao (Sp6), Jingmen(GB25), Yanglingquan (GB34) andXuanzhong (GB39) acupoints, while it was applied in the midline on Guanyuan (CV4) andMingmen (GV4) acupoints. Each acupoint was irradiated for 60 sec, with total duration of 20 min, wave length of 905 nm, average radiant power output of 12 mW, energy density of 2 J/cm2, pulse radiation of 200 ms and pulse frequency of 5000 Hz
  Arms: Drug treatment + laser acupuncture group

SUMMARY:
Sixty-eight postmenopausal women diagnosed with osteoporosis aged between 50 and 60 years were randomly allocated to one of two equal sets. The drug treatment group received calcium and vitamin D3 supplement daily for 12 weeks. While the drug/laser acupuncture group received laser acupuncture therapy for 20 minutes per session 3 times weekly, in addition to the same calcium and vitamin D3 supplement.

DETAILED DESCRIPTION:
Sixty-eight postmenopausal women diagnosed with osteoporosis were recruited from the outpatient clinic of obstetrics and gynaecology department, faculty of physical therapy, Cairo University. Women were enrolled and assessed for their eligibility to participate in the study. Inclusion criteria were: age between 50 and 60 years and the body mass index (BMI) between 25 and 35 Kg/m2. Multiparas with parity of 5 or more were included. They had decreased forearm BMD with T score of DEXA less than or equal to -2.5 and wrist pain with visual analogue scale (VAS) ≥ 3. They all have natural menopause for at least four years. They all were medically stable. Participants were excluded if they had history of bone disease, renal, liver, endocrinal or parathyroid disorders, cardiac affection, using a pacemaker or taking any drugs which may affect bone metabolism.

Each participant was informed about the study's nature, objective and usefulness, as well as her right to decline or leave the study at any time, and the confidentiality of any information gathered. A computer-based randomization program was used to randomize participants into two equal groups (Drug treatment Group and Drug treatment + LA Group). Drug treatment group (group A) included 34 postmenopausal women who only received oral calcium and vitamin D3 supplement (Calcium D3F® (Arab Company for Pharmaceutical& medicinal plants (MEPACO-MEDIFOOD, EGPYT). Each tablet contains 1000 mg of natural calcium carbonate, 1000 IU vitamin D3 (0.025 mg) and 0.25 mg Sodium Fluoride. They received 1 tablet once daily for 12 weeks. Drug treatment + laser acupuncture group (group B) included of 34 postmenopausal women who received laser acupuncture therapy in addition to the same calcium and vitamin D3 supplement for 12 weeks.

Each woman in group (B) received 3 sessions per week of laser acupuncture, for 12 weeks. The patient was in crock lying for stimulation of acupoints in abdomen and lower limbs then asked to be in side lying for stimulation of acupoints in the back. After disinfection of the skin and careful localization of the acupoints, low level laser therapy (LLLT) (model: Lis 1050, SN: EM 13481014, manufactured by EME srl, Italy) was applied bilaterally on Dazhu (BL 11), Ganshu(BL 18), Pishu (BL20), Shenshu (BL23), Zusanli (ST 36), Sanyinjiao (Sp6), Jingmen(GB25), Yanglingquan (GB34) andXuanzhong (GB39) acupoints, while it was applied in the midline on Guanyuan (CV4) andMingmen (GV4) acupoints. Each acupoint was irradiated for 60 sec, with total duration of 20 min, wave length of 905 nm, average radiant power output of 12 mW, energy density of 2 J/cm2, pulse radiation of 200 ms and pulse frequency of 5000 Hz

ELIGIBILITY:
Inclusion Criteria

* age between 50 and 60 years
* body mass index (BMI) between 25 and 35 Kg/m2.
* Multiparas with a parity of 5 or more were included.
* They had decreased forearm BMD with T score of DEXA less than or equal to -2.5 wrist pain with visual analogue scale (VAS) ≥ 3
* natural menopause for at least four years

Exclusion Criteria:

* history of bone disease, renal, liver, endocrinal or parathyroid disorders, cardiac affection,
* using a pacemaker
* taking any drugs which may affect bone metabolism

Ages: 50 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 68 (Actual)
Dates: Start 2021-07-11 (Actual); Primary Completion 2022-06-05 (Actual); Study Completion 2022-08-06 (Actual)

PRIMARY OUTCOMES:
Bone mineral density | 12 weeks after theray
  T-score of Forearm bone mineral density that was evaluated by dual energy X-ray absorptiometry
Pain Visual analogue score | 12 weeks after theray
  It is a 10-cm horizontal line on which a mark between the extremes of "no pain at all" and "worst agony conceivable" was used to reflect the patient's level of discomfort.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Maged, Principal Investigator — Cairo University
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

REFERENCES:
- [Derived] Hassan ES, Maged AM, Kotb A, Fouad M, El-Nassery N, Kamal WM. Effect of laser acupuncture on pain and density of bone in osteoporotic postmenopausal women: a randomized controlled trial. Menopause. 2023 May 1;30(5):545-550. doi: 10.1097/GME.0000000000002166. Epub 2023 Mar 20. PMID 36944142